CLINICAL TRIAL: NCT00574847
Title: Responses of Myocardial Ischemia to Escitalopram Treatment (REMIT Trial)
Brief Title: Responses of Myocardial Ischemia to Escitalopram Treatment
Acronym: REMIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00009555; R01HL085704-01 (NIH); 8640-07-8R1ER (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Ischemia
Keywords: ischemic heart disease; mental stress-induced myocardial ischemia; escitalopram
MeSH Terms: conditions — Myocardial Ischemia | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Experimental): Escitalopram treatment
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Dosage will range from 5 mg to 20 mg once a day for the duration of the study (6 weeks). Tablets are in 5 mg or 10 mg form, depending upon the dosage the patient is prescribed.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — Placebo dosage will range from 5 mg to 20 mg once a day for the duration of the study (6 weeks). Tablets are in 5 mg or 10 mg form, depending upon the dosage the patient is prescribed.
  Arms: Placebo

SUMMARY:
Depression is commonly seen in patients with cardiovascular disorders. In recent studies it has been shown that mild to moderate depression symptoms were associated with increased likelihood of mental stress-induced myocardial ischemia (MSIMI), which is a risk factor of poor cardiac outcome. In this project, the investigators aim to assess the treatment of mental stress-induced myocardial ischemia in ischemic heart disease patients with mild to moderate depressive symptoms. This study is a six-week double-blind placebo controlled study to examine the effects of escitalopram on mental stress-induced myocardial ischemia. This study will look to show that patients with ischemic heart disease who are treated with escitalopram will exhibit a significant improvement of MSIMI at the end of week 6 compared to patients receiving placebo.

DETAILED DESCRIPTION:
The goals of this project are to investigate the response of mental stress-induced myocardial ischemia (MSIMI) to escitalopram, a selective serotonin reuptake inhibitor (SSRI); to determine whether MSIMI will be reduced by the treatment, and whether the modification of MSIMI is related to improvement of depression symptoms, and/or the reduction of platelet aggregation, and/or the reduction of cardiovascular reactivity. This is a randomized study using escitalopram versus placebo for stable ischemic heart disease patients with MSIMI. This study will also explore the role of platelet activity in occurrence with MSIMI and other characteristics of MSIMI, such as systolic and diastolic function of the left ventricle during mental stress testing as compared to exercise testing.

The stress testing will be conducted at the Duke Cardiology Diagnostic Unit Laboratory. Following a 20-minute calibration-rest period, participants will be asked to complete a series of 3 mental stress tasks. There are 3 mental stress tasks to be used for this study, i.e., (1) Mental arithmetic: during this test, patients will be asked to perform a series of serial subtractions beginning at a given number which will be different for each repeated test and will be chosen by the tester from a fixed list of various numbers, with encouragement to perform calculations as quickly as possible; (2) Public speaking with anger recall: during this test, patients will be asked to give a speech on a recent situation in which they experienced anger to an audience of observers (two to three) after 1 minute of preparation. Prior to the speech, subjects are told that their speech will be evaluated on their description of the situation, as to what happened, what they thought, felt, what they did, and what happened as a result. If they run out of things to say, the research tech will prompt them with questions to elicit more content until the three minutes are up; (3) Mirror trace: during this test, patients will be asked to outline, as quickly as possible, a star from its reflection in a mirror. Each task will last 3 minutes and there will be a 6-minute rest period between tasks.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or greater, less than 90
* Stable ischemic heart disease

Exclusion Criteria:

* Recent myocardial infarction, coronary artery bypass graft surgery, or other revascularization procedures (less than 3 months ago)
* Left ventricular ejection fraction(LVEF) < 15% measured by echocardiography, radionuclide ventriculography (RNV), or cardiac catheterization
* Life threatening arrhythmia or arrhythmia interrupting the interpretation of ischemia
* Unable to withdraw from anti-anginal medications during ischemic assessment phase
* Unable to perform exercise testing
* Pregnancy
* Current or previous history of bipolar disorder, cyclothymia, schizophrenia, schizoaffective or schizophreniform disorder, or other psychotic disorders
* Active suicidal ideation
* Current substance abuse or history of substance abuse in the previous 6 months
* Significant cardiac, pulmonary, metabolic, renal, hepatic disease, or malignancy, interfering with patient's participation in this study
* Seizure (history and/or present) with/without treatment
* Currently taking antidepressants that cannot be discontinued

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Jiang W, Velazquez EJ, Samad Z, Kuchibhatla M, Martsberger C, Rogers J, Williams R, Kuhn C, Ortel TL, Becker RC, Pristera N, Krishnan R, O'Connor CM. Responses of mental stress-induced myocardial ischemia to escitalopram treatment: background, design, and method for the Responses of Mental Stress Induced Myocardial Ischemia to Escitalopram Treatment trial. Am Heart J. 2012 Jan;163(1):20-6. doi: 10.1016/j.ahj.2011.09.018. Epub 2011 Nov 14. PMID 22172432
- [Derived] Samad Z, Boyle S, Ersboll M, Vora AN, Zhang Y, Becker RC, Williams R, Kuhn C, Ortel TL, Rogers JG, O'Connor CM, Velazquez EJ, Jiang W; REMIT Investigators. Sex differences in platelet reactivity and cardiovascular and psychological response to mental stress in patients with stable ischemic heart disease: insights from the REMIT study. J Am Coll Cardiol. 2014 Oct 21;64(16):1669-78. doi: 10.1016/j.jacc.2014.04.087. PMID 25323254
- [Derived] Ersboll M, Al Enezi F, Samad Z, Sedberry B, Boyle SH, O'Connor C, Jiang W, Velazquez EJ; REMIT Investigators. Impaired resting myocardial annular velocities are independently associated with mental stress-induced ischemia in coronary heart disease. JACC Cardiovasc Imaging. 2014 Apr;7(4):351-61. doi: 10.1016/j.jcmg.2013.10.014. Epub 2014 Mar 13. PMID 24631512
- [Derived] Boyle SH, Samad Z, Becker RC, Williams R, Kuhn C, Ortel TL, Kuchibhatla M, Prybol K, Rogers J, O'Connor C, Velazquez EJ, Jiang W. Depressive symptoms and mental stress-induced myocardial ischemia in patients with coronary heart disease. Psychosom Med. 2013 Nov-Dec;75(9):822-31. doi: 10.1097/PSY.0b013e3182a893ae. Epub 2013 Oct 25. PMID 24163385
- [Derived] Jiang W, Velazquez EJ, Kuchibhatla M, Samad Z, Boyle SH, Kuhn C, Becker RC, Ortel TL, Williams RB, Rogers JG, O'Connor C. Effect of escitalopram on mental stress-induced myocardial ischemia: results of the REMIT trial. JAMA. 2013 May 22;309(20):2139-49. doi: 10.1001/jama.2013.5566. PMID 23695483
- [Derived] Jiang W, Samad Z, Boyle S, Becker RC, Williams R, Kuhn C, Ortel TL, Rogers J, Kuchibhatla M, O'Connor C, Velazquez EJ. Prevalence and clinical characteristics of mental stress-induced myocardial ischemia in patients with coronary heart disease. J Am Coll Cardiol. 2013 Feb 19;61(7):714-22. doi: 10.1016/j.jacc.2012.11.037. PMID 23410543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We screened all patients with Coronary Heart Disease (CHD) who visited Duke cardiology clinics. Patients 21 years or older were eligible to participate if they had CHD, as documented by angiographic findings of coronary artery stenosis of 70% or greater, history of MI, or history of cardiac revascularization.
Pre-assignment Details: 25527 underwent initial screening. 22833 excluded due to reasons including no CHD, atrial fibrillation/arrhythmia, psychiatric disorder, and LVEF less than 30%. 2294 did not provide consent. 65 excluded due to medical conditions. 203 excluded due to no MSIMI or inability to undergo mental stress testing. 5 more declined to undergo randomization.
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 64 | 63
Completed | 56 | 56
Not Completed | 8 | 7
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Did not receive medication (declined) | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.3) | 61.4 (11.5) | 64.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 53 | 48 | 101
History of Depression [Number; unit: participants] | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Absence of Mental Stress-induced Myocardial Ischemia (MSIMI) During the 3 Mental Stressors
Description: MSIMI is defined by the following: compared to rest, 1) any development of new abnormal wall motion; 2) reduction of LVEF 8% and/or; 3) deviation (depression or elevation) of ST-segment of ECG in 2 or more leads lasting for 3 consecutive beats, occurring during at least one of the 3 mental stress tasks.
Time Frame: Week 6
Population: Intent-to-treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 64 | 63
percentage of participants | 34.2 [31.6 to 36.8] | 17.5 [15.4 to 19.6]

2. Secondary Outcome: Mental Stress Induced Change of Systolic Blood Pressure
Description: Blood pressure will be measured the last 3 minutes of the 20 minute calibration period (resting), every minute during the 3 minutes mental stress testing, the last 3 minutes of the 6 minute rest periods between mental stress testing, and every minute during and after the physical stress testing with an automatic oscillometric blood pressure monitor (Quinton Electronics). Mental Stress Induced Change of Systolic Blood Pressure will be calculated by taking the mean of the mental stress systolic blood pressure measurements minus the resting Systolic blood pressure. End point values adjusted for baseline values age and sex.
Time Frame: Baseline, week 6
Population: ITT, 9 subjects excluded from analysis due to missing data.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 62 | 56
mm Hg | 19.3 [16.7 to 22.0] | 23.6 [20.8 to 26.4]

3. Secondary Outcome: Mental Stress Induced Change of Diastolic Blood Pressure
Description: Blood pressure will be measured the last 3 minutes of the 20 minute calibration period (resting), every minute during the 3 minutes mental stress testing, the last 3 minutes of the 6 minute rest periods between mental stress testing, and every minute during and after the physical stress testing with an automatic oscillometric blood pressure monitor (Quinton Electronics). Mental Stress Induced Change of Diastolic Blood Pressure will be calculated by taking the mean of the mental stress Diastolic blood pressure measurements minus the resting Diastolic blood pressure. End point values adjusted for baseline values age and sex.
Time Frame: Baseline, week 6
Population: ITT, 9 subjects excluded from the analysis due to missing data.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 62 | 56
mm Hg | 11.4 [9.5 to 13.4] | 12.2 [10.1 to 14.2]

4. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Baseline to week 6
Measure: Number; unit: percentage of participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 64 | 63
percentage of participants | 71.9 | 44.4

5. Secondary Outcome: Beck Depression Inventory
Description: The Beck Depression Inventory II (BDI-II) is a 21 question, self-administered measure of depressive symptoms. Score range, 0 to 63 (higher score=greater severity of depressive symptoms). End point values adjusted for baseline values age and sex.
Time Frame: 6 week
Population: ITT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 64 | 63
units on a scale | 7.4 [6.3 to 8.6] | 7.0 [5.8 to 8.2]

6. Secondary Outcome: Mental Stress Induced Change in Heart Rate
Description: A standard 12-lead Electrocardiograph (ECG) will be recorded at 1-minute intervals during the last 3 minutes of each rest period, the 3 minutes of the mental stress testing, and during exercise testing. Heart rate will be determined from the ECGs.
  Mental Stress Induced Change in heart rate will be calculated by taking the mean of the mental stress heart rate measurements minus the resting heart rate measurements. End point values adjusted for baseline values age and sex.
Time Frame: baseline, 6 weeks
Population: ITT, 10 subjects excluded from analysis due to missing data.
Measure: Mean (95% Confidence Interval); unit: beats/minute
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 61 | 56
beats/minute | 6.34 [5.0 to 7.7] | 9.1 [7.8 to 10.5]

7. Secondary Outcome: 5HTT, Serotonin Transporter Protein
Description: End point values adjusted for baseline values age and sex.
Time Frame: week 6
Population: ITT, 29 subjects excluded from analysis due to missing data.
Measure: Mean (95% Confidence Interval); unit: fmol/mg
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 48 | 50
fmol/mg | 139.7 [126.1 to 153.4] | 160.4 [147.0 to 173.7]

8. Secondary Outcome: Platelet Serotonin Binding Affinity Kd_100
Description: End point values adjusted for baseline values age and sex.
Time Frame: 6 weeks
Population: ITT, 27 subjects were excluded from analysis due to missing data.
Measure: Mean (95% Confidence Interval); unit: nM
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 50 | 50
nM | 4202.4 [3328.6 to 5076.2] | 210.1 [0.0 to 1083.9]

9. Secondary Outcome: Perceived Stress Scale
Description: Score range, 10 to 50 (higher score = greater levels of perceived stress). End point values adjusted for baseline values age and sex.
Time Frame: 6 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 64 | 63
units on a scale | 21.4 [20.3 to 22.5] | 21.8 [20.6 to 22.9]

10. Secondary Outcome: Cook-Medley Hostility (Ho) Scale
Description: Score ranges: hostility, 0 to 27 (higher score=greater levels of hostility)/ End point values adjusted for baseline values age and sex.
Time Frame: 6 weeks
Population: ITT, 1 subject excluded from analysis due to missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 64 | 62
units on a scale | 9.9 [9.1 to 10.7] | 10.3 [9.5 to 11.1]

11. Secondary Outcome: Cook-Medley Hostility (Ho) Hostile Affect Sub-scale
Description: hostile affect, 0 to 5 (higher score=greater levels of hostile affect). End point values adjusted for baseline values age and sex.
Time Frame: 6 weeks
Population: ITT, 1 subject excluded from analysis due to missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 64 | 62
units on a scale | 1.6 [1.3 to 1.8] | 1.8 [1.6 to 2.1]

12. Secondary Outcome: Spielberger State-Trait Anxiety Inventory Scales (STAI)
Description: STAI measures anxiety. The questionnaire asks the patients how they feel and allows them to respond on a frequency scale that ranges from 1(not at all) to 4(almost always/very much so). Scores range from 20-80 and the higher the score the greater the anxiety level. This applies to both the Trait and State scales. End point values adjusted for baseline values age and sex.
Time Frame: 6 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 64 | 63
units on a scale
  Trait | 31.2 [29.7 to 32.6] | 32.0 [30.5 to 33.4]
  State | 27.9 [26.4 to 29.4] | 29.5 [28.0 to 31.1]

13. Secondary Outcome: Exercise Stressed-induced Myocardial Ischemia (ESIMI)
Description: End point values adjusted for baseline values age and sex.
Time Frame: 6 week
Population: ITT, 7 subject excluded from analysis due to missing data.
Measure: Number (95% Confidence Interval); unit: percentage of change
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 59 | 61
percentage of change | 45.8 [36.6 to 55.0] | 52.5 [43.3 to 61.8]

14. Primary Outcome: Percentage of Participants With Overall Mental Stress-induced Myocardial Ischemia (MSIMI)
Description: as for outcome 1
Time Frame: week 6
Population: Subjects who completed.
Measure: Number; unit: percentage of participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 56 | 56
percentage of participants | 66.1 | 83.9

ADVERSE EVENTS:
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 3/64 | 1/63
Other Adverse Events (participants affected / at risk) | 46/64 | 28/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=64) | Placebo (N=63)
Confusion, Hallucination (Nervous system disorders) | 1 | 0
Death (Cardiac disorders) | 1 | 0
unstable angina (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=64) | Placebo (N=63)
fatigue (General disorders) | 19 | 9
burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
CNS symptom (Nervous system disorders) | 17 | 13
constipation (Gastrointestinal disorders) | 18 | 11
cramping in legs (Musculoskeletal and connective tissue disorders) | 3 | 2
irregular heartbeat (Cardiac disorders) | 0 | 2
sexual dysfunction (Reproductive system and breast disorders) | 10 | 4
sinusitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes